CLINICAL TRIAL: NCT01770574
Title: Structural HATCP Graft vs Tricortical Iliac Crest Autograft in Paediatric Calcaneal Lengthening Osteotomies: Interim Results From a Randomised Controlled Noninferiority Study
Brief Title: New Bone Grafting Technique in Paediatric Foot Surgery. Validation of Outcome Measures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim results showed that the HATCP material was not non-inferior to the AUTO graft.
Sponsor: University of Aarhus (Other)
Collaborators: Ceramisys Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-250-12; Interventional (Other: Videnskabsetisk Komité)
Record Dates: First submitted 2012-09-26; First posted 2013-01-18 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2016-07

CONDITIONS: Pes Planovalgus
Keywords: calcaneal lengthening; calcium ceramics; noninferiority; radiostereometric analysis
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ReproBone (Experimental): calcaneal lengthening
  Interventions: Device: ReproBone; Procedure: calcaneal lengthening
- Autologous bone graft (Active Comparator): calcaneal lengthening
  Interventions: Procedure: calcaneal lengthening

INTERVENTIONS:
Device: ReproBone — Artificial bone graft is inserted as a wedge in the calcaneal lengthening osteotomy
  Other Names: Hydroxy-apatite-tricalcium-phosphate
  Arms: ReproBone
Procedure: calcaneal lengthening — Autologous bone graft is harvested from the iliac crest and inserted as a wedge in the calcaneal lengthening osteotomy
  Other Names: Autologous bone graft

SUMMARY:
The purpose of this study is to determine whether structural calcium ceramic bone graft substitute (ReproBone™) is non-inferior compared to autologous tricortical iliac crest bone graft in lateral calcaneal lengthening osteotomies in pediatric patients and reduces postoperative pain.

To groups of patients (age 5-16) will be compared. One group randomized to autologous bone graft and the other group randomized to calcium ceramic.

The evaluation will be based on radiostereometric analysis, pedobarography, Patient reported outcome assessment (Oxford Ankle Foot Questionnaire), and pain (measured by visual analog scale and numerical range scale).

DETAILED DESCRIPTION:
Study C: HA-β TCP (ReproBone™) vs. autologous tricortical iliac crest bone graft in a calcaneal lengthening osteotomy in children with pes planovalgus. A clinical randomized controlled non-inferiority study with 12 months of follow-up.

Purpose. To investigate the clinical and radiographic findings of a calcaneal lengthening osteotomy by comparing autologous bonegraft and HA-β-TCP graft in a group of children with hindfoot valgus deformities. The primary outcome measure the stability of the osteotomy measured by migrations in the x-translation by RSA.

Design. Prospective, randomized controlled non-inferiority study.

Randomization: Children who fulfill the criteria for inclusion together with their parents/guardian receive information about the project. The patients are randomized to respectively HA-ß-TCP and iliac crest bone graft.

Surgical procedure: Calcaneal lengthening osteotomy is performed between the anterior and middle facet of the subtalar joint. The corticalis of the calcaneus is bilaterally cut through. The planovalgus deformity is corrected and with a graft matching the wedged osteotomy is inserted. Tantalum balls are inserted into calcaneus on each side of the osteotomy and in cuboideum. Postoperative pain treatment consist of a tibial nerve catheter which is used the first 24 hours. Patients in whom graft is harvested from the iliac crest get local infiltration analgesics accordingly to a standardized procedure. The pain is registered by the use of a visual analog scale (VAS, NRS, faces scale) a 3, 8 and 12 hours postoperative. The amounts of used analgesics are registered. The stability of the osteotomy is assessed by radiostereometric assay (RSA) at the following time points: Baseline (first/second postoperative day) after 6 weeks, 8 weeks, 6 months and 12 months.

Power and significance: The primary parameter is stability of the osteotomy, measured as x-translations by the RSA software. We used continuous non-inferiority sample size calculations. With alpha 0.05 and power 0.9, non-inferiority limit 2 mm and sd 1.5 mm we estimated the sample size to 10 patients in each group. To secure against drop-out, we plan to include 15 patients in each group.

For ethical considerations an interim analysis was planned when 10 patients completed 6 months RSA follow-up. Primary outcome was compression of the osteotomy. We used a 99.8% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 5-16 years with symptomatic planovalgus deformity admitted to the Department of Children's Orthopaedics, Aarhus University Hospital during the period 2012 to 2016. The surgical procedure is performed in about 10 children a year.

Pain and/or callosities. Informed written consent from the child custody/guardianship. Ambulatory function No severe cognitive deficits

Exclusion Criteria:

Reoperation will exclude patients from further follow-up

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2013-02; Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-10 (Actual)

PRIMARY OUTCOMES:
Radiostereometric Analysis (RSA) of the calcaneal lengthening osteotomy | Postoperative, 6 weeks, 8 weeks, 6 months, 12 months
  RSA examinations will be performed at baseline (first/second postoperative day), after 6 weeks, 8 weeks, 6 months and 12 months. Aim: To assess stability of the osteotomy and any micro motion in the neighbouring calcaneal-cuboid joint.

SECONDARY OUTCOMES:
General Pain | The first 24 hrs after surgery
  Pain will be assessed as general pain, by VAS/NRS/faces scaling at baseline (pre-op), 3 hrs, 5 hrs, 8 hrs, 12 hrs after surgery. Although minor changes in the specific time points can occur if the child is sleeping, since it would be unethical to wake them up.

OTHER OUTCOMES:
Pedobarography | preoperative, 6 months, 12 months
  Pedobarography: The investigators use a pressure plate from Tekscan. The pressure of the patients feet is measures during stance and walking.
OxAFQ | preoperative, 6 months, 12 months
  health related quality of life in children with foot/ankle issues

CONTACTS AND LOCATIONS:
Overall Officials: Bjarne Møller-Madsen, DMSc, Prof, Study Director — Department of Children's Orthopaedics Aarhus University Hospital; Polina Martinkevich, PhD-student, Principal Investigator — Department of Children's Orthopaedics Aarhus University Hospital; Ole Rahbek, Assoc prof PhD MD, Study Chair — Department of Children's Orthopaedics, Aarhus University Hospital; Martin Gottliebsen, MD PhD-stud, Study Chair — Department of Children's Orthopaedics, Aarhus University Hospital; Maiken Stilling, MD, PhD, Study Chair — Department of Orthopaedics, Aarhus University Hospital; Line Kjeldgaard Pedersen, MD, PhD, Study Chair — Department of Children's Orthopaedics, Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark